CLINICAL TRIAL: NCT07338773
Title: Comparison of the Effects of Intraosseous and Intravenous Vancomycin Prophylaxis on Surgical Site Infections and Clinical Outcomes After Diabetic Foot Amputation: A Randomized Controlled Trial
Brief Title: Intraosseous vs. Intravenous Vancomycin Prophylaxis for Diabetic Foot Amputations: A Randomized Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Lezgin Mert, Orthopaedic surgeon, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-96317027-514.10-285164594
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Disease; Diabetic Foot Infection; Diabetic Amputation Foot Wound
Keywords: DIABETIC FOOT, VANCOMYCIN INTRAOSSEOUS, AMPUTATION
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE, RANDOMIZED, PARALLEL-ASSIGNMENT, CONTROLLED CLINICAL TRIAL. PATIENTS ARE RANDOMLY ASSIGNED TO EITHER THE INTRAOSSEOUS (IO) VANCOMYCIN GROUP OR THE INTRAVENOUS (IV) VANCOMYCIN GROUP IN A 1:1 RATIO.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraosseous Vancomycin (Experimental): 500 mg Vancomycin hydrochloride dissolved in of %0.9 NaCl, administered directly into the intramedullary space.
  Interventions: Drug: Intraosseous Vancomycin
- Intravenous Vancomycin (Active Comparator): 500 mg Vancomycin hydrochloride administered via peripheral intravenous infusion
  Interventions: Drug: Intravenous Vancomycin

INTERVENTIONS:
Drug: Intraosseous Vancomycin — A single dose of 500 mg Vancomycin is administered into the bone marrow (intraosseous route) to achieve high local tissue concentrations at the surgical site.
  Arms: Intraosseous Vancomycin
Drug: Intravenous Vancomycin — A single dose of 500 mg Vancomycin is administered via systemic intravenous infusion for standard prophylactic care.
  Arms: Intravenous Vancomycin

SUMMARY:
he purpose of this study is to compare the effects of two different ways of giving the antibiotic vancomycin to prevent infections in patients undergoing amputation due to diabetic foot infection. Patients with diabetes often have poor blood circulation in their legs, which may prevent standard intravenous (IV) antibiotics from reaching the surgical site in high enough concentrations.

This study compares:

Intraosseous (IO) Administration: Giving the antibiotic directly into the bone at the amputation site during surgery.

Intravenous (IV) Administration: Giving the antibiotic through a standard vein infusion before surgery.

The researchers want to find out if the intraosseous method:

Reduces the rate of surgical site infections compared to the standard IV method.

Causes fewer changes in kidney function (measured by serum creatinine levels). Decreases the need for additional surgeries (reoperations) within 90 days. Patients will be randomly assigned to either the IO or IV group and will be followed for up to 90 days to evaluate their recovery and clinical outcomes

DETAILED DESCRIPTION:
DETAILED DESCRIPTION THE SURGICAL MANAGEMENT OF DIABETIC FOOT INFECTIONS IS OFTEN COMPLICATED BY PERIPHERAL VASCULAR DISEASE, WHICH SIGNIFICANTLY IMPAIRS THE DELIVERY OF SYSTEMIC PROPHYLACTIC ANTIBIOTICS TO THE INFECTED OR ISCHEMIC EXTREMITY. THIS PROSPECTIVE, RANDOMIZED, CONTROLLED STUDY INVESTIGATES WHETHER INTRAOSSEOUS (IO) ADMINISTRATION OF VANCOMYCIN PROVIDES A SUPERIOR CLINICAL OUTCOME BY DELIVERING HIGHER LOCAL TISSUE CONCENTRATIONS COMPARED TO TRADITIONAL INTRAVENOUS (IV) ADMINISTRATION.

STUDY RATIONALE AND HYPOTHESIS: PREVIOUS STUDIES IN TOTAL KNEE ARTHROPLASTY HAVE SHOWN THAT IO ADMINISTRATION INCREASES LOCAL ANTIBIOTIC TISSUE CONCENTRATION WHILE REDUCING SYSTEMIC LEVELS. DUE TO PERIPHERAL VASCULAR DISEASE IN DIABETIC FOOT PATIENTS, WE BELIEVE THAT SYSTEMICALLY ADMINISTERED VANCOMYCIN (IV) WILL REACH LOWER CONCENTRATIONS AT THE SURGICAL SITE. WE HYPOTHESIZE THAT INTRAOSSEOUS VANCOMYCIN WILL ACHIEVE SIGNIFICANTLY HIGHER DRUG LEVELS IN THE AMPUTATION STUMP AREA, REDUCE THE RATE OF SURGICAL SITE INFECTIONS (SSI), RESULT IN SMALLER INCREASES IN SERUM CREATININE LEVELS DUE TO LOWER SYSTEMIC EXPOSURE, AND DECREASE THE NECESSITY FOR REOPERATION (RTOR) IN PATIENTS UNDERGOING TRANSTIBIAL AMPUTATION.

METHODOLOGY AND INTERVENTIONS: PATIENTS ARE RANDOMIZED IN A 1:1 RATIO INTO TWO TREATMENT ARMS:

IO GROUP: DURING THE AMPUTATION PROCEDURE, 500 MG OF VANCOMYCIN IS ADMINISTERED VIA THE INTRAOSSEOUS ROUTE DIRECTLY AT THE AMPUTATION SITE.

IV GROUP: PATIENTS RECEIVE 500 MG OF VANCOMYCIN INTRAVENOUSLY 15-30 MINUTES PRIOR TO THE SURGICAL INCISION.

PHARMACOKINETIC EVALUATION (PRIMARY FOCUS): VANCOMYCIN CONCENTRATIONS WILL BE MEASURED FROM BOTH THE STUMP SITE (LOCAL TISSUE) AND SYSTEMIC CIRCULATION (PERIPHERAL BLOOD) TO COMPARE THE DISTRIBUTION AND CONCENTRATION GRADIENTS OF THE DRUG BETWEEN THE TWO ADMINISTRATION ROUTES. SAMPLES WILL BE COLLECTED INTRAOPERATIVELY TO DETERMINE IF THE IO ROUTE BYPASSES VASCULAR INSUFFICIENCY.

FOLLOW-UP AND OUTCOME EVALUATION: PATIENTS WILL BE FOLLOWED POSTOPERATIVELY ON DAYS 1,2,3,7 AND 30 FOR CLINICAL OUTCOMES ACCORDING TO CDC CRITERIA. SECONDARY OUTCOMES, INCLUDING SERUM CREATININE LEVELS TO MONITOR RENAL SAFETY AND REOPERATION RATES (REVISION AMPUTATION, DEBRIDEMENT), WILL BE TRACKED FOR UP TO 90 DAYS. MULTIVARIATE LOGISTIC REGRESSION WILL BE USED TO ADJUST FOR CONFOUNDING FACTORS SUCH AS AGE, GENDER, AND HBA1C LEVELS.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS AGED 18 YEARS AND OLDER. DIAGNOSED WITH TYPE 1 OR TYPE 2 DIABETES MELLITUS. SCHEDULED FOR TRANSTIBIAL (BELOW-KNEE) AMPUTATION DUE TO DIABETIC FOOT INFECTION.

WILLING AND ABLE TO PROVIDE WRITTEN INFORMED CONSENT.

Exclusion Criteria:

KNOWN ALLERGY OR HYPERSENSITIVITY TO VANCOMYCIN.

PRE-EXISTING RENAL INSUFFICIENCY (BASELINE SERUM CREATININE > 2.0 MG/DL OR GFR < 30 ML/MIN).

PREGNANCY OR BREASTFEEDING.

PREVIOUS SURGICAL INTERVENTION OR AMPUTATION ON THE SAME EXTREMITY.

BODY MASS INDEX (BMI) OVER 35.

CONTRAINDICATION TO STANDARD PROPHYLACTIC ANTIBIOTICS.

INABILITY TO LOCALIZE THE TIBIAL TUBERCLE FOR INTRAOSSEOUS INFUSION.

IMMUNOCOMPROMISED STATUS (HIV, HEPATITIS C, END-STAGE RENAL DISEASE, DIALYSIS, ACTIVE CHEMOTHERAPY OR RADIOTHERAPY).

USE OF IMMUNOSUPPRESSIVE DRUGS WITHIN THE LAST 6 MONTHS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
LOCAL AND SYSTEMIC VANCOMYCIN CONCENTRATIONS | NTRAOPERATIVE (MEASURED DURING SURGERY, APPROXIMATELY 15-30 MINUTES AFTER DRUG ADMINISTRATION).
  COMPARISON OF VANCOMYCIN CONCENTRATIONS (MCG/ML) MEASURED FROM THE SURGICAL SITE (LOCAL STUMP AREA) AND THE SYSTEMIC CIRCULATION (PERIPHERAL BLOOD). THE GOAL IS TO EVALUATE THE PHARMACOKINETIC EFFICIENCY OF INTRAOSSEOUS (IO) ADMINISTRATION VERSUS INTRAVENOUS (IV) ADMINISTRATION IN REACHING TARGET LEVELS AT THE AMPUTATION SITE IN PATIENTS WITH PERIPHERAL VASCULAR DISEASE.

SECONDARY OUTCOMES:
REOPERATION RATE (RTOR) | UP TO 30 DAYS POSTOPERATIVELY.
  ECESSITY FOR ADDITIONAL SURGICAL INTERVENTION, SUCH AS REVISION AMPUTATION OR DEBRIDEMENT.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam ve Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the final article, after de-identification (including text, tables, figures, and appendices), will be made available to researchers whose proposed use of the data has been approved by a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 2 months and ending 12 months after article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to achieve the objectives in the approved proposal. Proposals should be directed to the corresponding author's email.

REFERENCES:
- [Result] Wininger AE, Gurusamy P, Sullivan TC, Serpelloni S, Taraballi F, Park KJ, Brown TS. Intraosseous Versus Intravenous Vancomycin in Tourniquetless Primary Total Knee Arthroplasty: A Randomized Trial. J Arthroplasty. 2024 Sep;39(9S2):S224-S228. doi: 10.1016/j.arth.2024.02.083. Epub 2024 Mar 8. PMID 38462143